CLINICAL TRIAL: NCT03837548
Title: A Phase 1 Double-Blind Crossover Comparative Study of Neurofeedback for the Treatment of Parkinson's Disease
Brief Title: A Study of Neurofeedback for the Treatment of Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18027-2; UMIN000032937 (Registry Identifier: University Hospital Medical Information Network Clinical Trials Registry (UMIN-CTR))
Record Dates: First submitted 2019-01-15; First posted 2019-02-12 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Magnetoencephalography; Neurofeedback
MeSH Terms: conditions — Parkinson Disease | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training with Neurofeedback (Experimental)
  Interventions: Other: Training with Neurofeedback
- The other Training with Neurofeedback (Experimental)
  Interventions: Other: The other Training with Neurofeedback

INTERVENTIONS:
Other: Training with Neurofeedback — Neurofeedback the brain activities by Magnetoencephalography
  Arms: Training with Neurofeedback
Other: The other Training with Neurofeedback — Neurofeedback the brain activities by Magnetoencephalography
  Arms: The other Training with Neurofeedback

SUMMARY:
This study aims to reveal relationship between brain activities and the symptoms of Parkinson disease when a neurofeedback training was applied for them.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with age more than 20
* Subjects obtained the consent
* Subjects with Parkinson disease and healthy subjects

Exclusion Criteria:

* The subjects who can not conduct the tasks
* Subjects with severe illness
* Subjects whom the experimenter think as in appropriate
* Subjects with implantable devices such as pacemaker

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Alteration of Brain Activities | At the time Immediately following the training
  measured by magnetoencephalography

SECONDARY OUTCOMES:
The raw score change from baseline in the Movement disorder society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part Ⅲ scores | At the time Immediately following the training
  MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The scales are now titled; (Part I) nonmotor experiences of daily living (13 items), (Part II) motor experiences of daily living (13 items), (Part III) motor examination (18 items), and (Part IV) motor complications (six items). Each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.
  The total score is the sum of the subscale scores for Part III and ranges from 0 (no disability) to 132 (total dependence).

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka University, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Izutsu N, Yanagisawa T, Fukuma R, Kishima H. Magnetoencephalographic neurofeedback training decreasesbeta-low-gammaphase-amplitude coupling of the motor cortex of healthy adults: a double-blinded randomized crossover feasibility study. J Neural Eng. 2023 May 9;20(3). doi: 10.1088/1741-2552/acd0d6. PMID 37105162